CLINICAL TRIAL: NCT01530191
Title: Factors Affectign Perioperative Outcomes After Surgery for Pelvic Organ Prolapse
Brief Title: Factors Affecting Perioperative Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: No subject accrual
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: shobeiridepression_10.18.11
Record Dates: First submitted 2012-01-19; First posted 2012-02-09 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: depression; anxiety; pelvic organ prolapse; POP
MeSH Terms: conditions — Pelvic Organ Prolapse; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Abdominal: - Participants undergoing surgeries with an abdominal approach will be given a Morphine PCA at a dose of 2mg every 10 minutes with a 12mg/hour lockout. They will also be given IV Toradol at 30mg every 6 hours as needed for a maximum of four doses.
- Vaginal: - Participants undergoing surgeries with a vaginal approach will be given hydrocodone/acetaminophen at a dose of 5/325 (1-2 tablets every four hours as needed), and provided with Ibuprofen 800mg every 8 hours as needed.

SUMMARY:
The specific aim of this study is to determine if pre-existing depression and anxiety affect perioperative outcomes measures patients undergoing surgery for pelvic organ prolapse.

* Hypothesis 1: Patients with depression will have increased analgesic use and longer hospital stays postoperatively
* Hypothesis 2: Patients with anxiety will have increased analgesic use and longer hospital stays postoperatively.

A secondary aim is to characterize the incidence and severity of depression and anxiety in patients scheduled to undergo surgery for pelvic organ prolapse.

DETAILED DESCRIPTION:
Objectives: The purpose of this study is to assess preoperative depression and anxiety in patients scheduled to undergo surgery for pelvic organ prolapse and to determine if pre-existing depression and anxiety will affect perioperative outcomes in this patient population.

Methodology: Patients from the University of Oklahoma Urogynecology clinics who have been scheduled to undergo surgery for pelvic organ prolapse will be invited to participate in this study. Informed consent will be obtained prior to study enrollment. Data obtained from a preoperative visit with each participant will include demographic information, medical and surgical histories, and a complete physical examination. After enrollment into the study, each participant will be started on a standardized dose of analgesics. The visual analog scale will be used to assess the level of pain at the surgical site and pain medications will be adjusted as necessary. Information regarding their postoperative course will be tracked, including any complications, use of pain medications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 21
* Scheduled to undergo surgery for the treatment of pelvic organ prolapse at the University of Oklahoma Health Sciences Center

Exclusion Criteria:

* Age < 21
* Inability to complete the written questionnaires
* Undergoing concurrent procedures for condition other than pelvic organ prolapse

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the University of Oklahoma Urogynecology clinics. Our catchment area includes OU Physicians clinic (private clinic) and Presbyterian Professional Building (resident clinic).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | 1 week
Analgesic use | 1 week
Length of hospital stay | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Mikio Nihira, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States